CLINICAL TRIAL: NCT03478865
Title: An Investigation of Vitamin A Palmitate Supplementation in Patients With Age-Related Macular Degeneration (and Without Reticular Pseudodrusen) and Delayed Dark Adaptation
Brief Title: Vitamin A Palmitate Supplementation in People With Age-Related Macular Degeneration (and Without Reticular Pseudodrusen) and Delayed Dark Adaptation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180067; 18-EI-0067
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-03

CONDITIONS: AMD
Keywords: Eye Examinations; Retinal Pigment Epithelium
MeSH Terms: interventions — retinol palmitate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants with age-related macular degeneration
  Interventions: Drug: Vitamin A palmitate

INTERVENTIONS:
Drug: Vitamin A palmitate — Provide vitamin A to participants with pre/post assessments of vision.

SUMMARY:
Background:

Age-related macular degeneration (AMD) is an eye disease. It is the leading cause of vision loss in people over 55 in the U.S. Changes in the eye can make it difficult for the eye to adjust to low light. This is known as dark adaptation. Identifying and watching the early to middle stages of AMD and changes in dark adaptation might help researchers develop new treatments to stop the disease before it becomes severe. Taking vitamin A might help improve vision in people with AMD.

Objectives:

To see if taking 16,000 IU of vitamin A per day improves vision in people with AMD. Also to improve understanding of AMD and associated dark adaptation.

Eligibility:

Adults ages 50 and older with AMD and normal liver function

Design:

Participants will be screened with:

Medical and eye disease history

Eye exam: The pupil will be dilated with eye drops. Pictures will be taken of the retina and the inside of the eye.

Including the screening visit, participants will have at least 5 visits. They will be about once a month over 6 months. Visits include:

Questions about eye problems in certain light

Eye exam

Blood and urine tests

Dark adaptation protocol: Participants will sit at a machine in a dark room. They will look into the machine and push a button when they see a light. This lasts 20-30 minutes.

Participants will take a vitamin A supplement by mouth once a day for 2 months. They will record when they take the pills in a diary.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to investigate the potential efficacy and safety of vitamin A palmitate dosing in improving dark adaptation in participants with age-related macular degeneration (AMD) and abnormal dark adaptation.

Study Population:

The first cohort consists of five participants with AMD who meet the eligibility criteria. The second cohort will consist of five participants with AMD who meet the eligibility criteria. Up to five additional participants may be accrued in the second cohort to account for participants who withdraw from the study prior to receiving one month of study supplementation for a reason unrelated to an adverse reaction. Up to 18 participants may be enrolled in this study.

Design:

This is a prospective, uncontrolled, single center, pilot study to investigate the potential efficacy and safety of vitamin A palmitate dosing in improving dark adaptation in participants with AMD and abnormal dark adaptation. Participants in the first cohort were instructed to take 16,000 IU of vitamin A palmitate daily for two months. Enrollment for Cohort 1 ended on May 24, 2019. Participants in the second cohort will be instructed to take 48,000 IU of vitamin A palmitate daily for one month. Participants in both cohorts will continue in the study for one month after ending Vitamin A supplementation. Participants in Cohort 1 may enroll into Cohort 2 as long as their last intake of vitamin A palmitate was greater than two months prior to their enrollment into Cohort 2.

Outcome Measures:

For each cohort, the primary outcome is the measurement of dark adaptation parameters (thresholds and kinetics) by the following: dark adaptation times as measured by the AdaptDx comparing before and after vitamin A palmitate supplementation and dark adaptation parameters as measured by the Medmont comparing before and after vitamin A palmitate supplementation. The primary outcome will be assessed at Month 2 in the first cohort and Month 1 in the second cohort. For both cohorts, the secondary outcomes include changes in low luminance visual acuity (LLVA) and changes in patient reported outcomes as measured by the low luminance questionnaire (LLQ). The secondary outcomes also include measurement of dark adaptation parameters (thresholds and kinetics) comparing baseline and one month after completing supplementation (Month 3 in Cohort 1 and Month 2 in Cohort 2).

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

* Participant must be 50 years of age or older.
* Participant must understand and sign the protocol s informed consent document.
* Any participant of childbearing potential must be willing to undergo urine pregnancy tests throughout the study.
* Any participant of childbearing potential and any participant able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse, or must agree to practice at least one acceptable method of contraception throughout the course of the study and for one week after study supplement discontinuation. Acceptable methods of contraception include:

  * Hormonal contraception (i.e. birth control pills, injected hormones, dermal patch or vaginal ring),
  * Intrauterine device,
  * Barrier methods (diaphragm, condom) with spermicide, or
  * Surgical sterilization (tubal ligation).
* Participants must agree to notify the study investigator or coordinator if any of their doctors initiate a new prescription medication during the course of this study.
* Participant must agree to not take greater than or equal to 8000 IU vitamin A palmitate outside the study supplementation.
* For supplementation eligibility, participant must have normal liver function as demonstrated by the Chemistry 20 panel, or have mild abnormalities not above grade 1 as defined by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE).

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present:

* Participant is in another investigational study and actively receiving study therapy.
* Participant is unable to comply with study procedures or follow-up visits.
* Participant is already taking vitamin A palmitate supplements greater than or equal to 8,000 IU.
* Participant has a history of vitamin A deficiency.
* Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
* Participant has a history of hepatitis or liver failure.
* Participant has chronic gastrointestinal disease.
* Participant will be excluded if the participant has serologic evidence of an active hepatitis infection.
* Participant was in Cohort 1 and took his/her last dose of vitamin A palmitate less than two months prior to enrolling in Cohort 2.

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

STUDY EYE INCLUSION CRITERIA:

* The eye must have a best-corrected ETDRS visual acuity score better than or equal to 20/80 (i.e., equal to or better than 54 letters).
* Participant must have at least one large druse.
* Abnormal dark adaptation, which is defined as having an Adapt Dx test with a RIT of 16 minutes or more at the screening visit. This is at least one standard deviation greater than the average normal RIT and includes room to account for variability in testing. If at any point during current testing or under a previous NEI protocol, a participant has exceeded the 40 minute test ceiling, they will have satisfied the inclusion criteria.

STUDY EYE EXCLUSION CRITERIA:

* Presence of advanced macular degeneration with central geographic atrophy or choroidal neovascularization.
* Presence of definite reticular pseudodrusen.
* An ocular condition is present (other than retinal vein occlusion) that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of major ocular surgery (e.g. cataract extraction, scleral buckle, any intraocular surgery, etc.) within three months prior to study entry.
* History of YAG (Yttrium-Aluminum Garnet) capsulotomy performed within two months prior to study entry.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pfau K, Jeffrey BG, Cukras CA. LOW-DOSE SUPPLEMENTATION WITH RETINOL IMPROVES RETINAL FUNCTION IN EYES WITH AGE-RELATED MACULAR DEGENERATION BUT WITHOUT RETICULAR PSEUDODRUSEN. Retina. 2023 Sep 1;43(9):1462-1471. doi: 10.1097/IAE.0000000000003840. PMID 37315571
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-EI-0067.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to eighteen (18) participants (8 participants in Cohort 1 and up to 10 participants in Cohort 2) with age-related macular degeneration (AMD) and abnormal dark adaptation may be enrolled. At the National Eye Institute, enrollment for Cohort 1 closed on May 24, 2019 and enrollment for Cohort 2 was suspended on August 31, 2023.
Pre-assignment Details: Participants met all inclusion criteria and none of the exclusion criteria for at least on eye as defined in the protocol. If both eyes met the eligibility criteria, the eye with the better visual acuity was chosen as the study eye. Participants enrolled after May 24, 2019 were enrolled into Cohort 2. All eligible participants underwent treatment starting at Baseline. The IP used in the study was vitamin A palmitate and was not anticipated to differentially treat participant eyes.
Groups:
- Cohort 1: Oral administration of vitamin A palmitate. Vitamin A palmitate: Participants in Cohort 1 were instructed to take 16,000 international unit of investigational product (IP) daily for two months. At Baseline and Month 1, a one month supply of IP was dispensed to the participant during the study visit. Participants were required to bring their bottles of IP to each appropriate visit for IP counts for compliance monitoring. Participants could complete participation in the study one month after IP supplementation (Month 3). At the conclusion of the study, participants were no longer eligible to receive IP under this protocol.
- Cohort 2: Oral administration of vitamin A palmitate. Vitamin A palmitate: Participants in Cohort 2 were instructed to take 48,000 international unit of investigational product (IP) daily for one month. Participants in Cohort 1 could enroll into Cohort 2 as long as their last intake of vitamin A palmitate was greater than two months prior to their enrollment into Cohort 2. At Baseline, a one month supply of IP was dispensed to the participant during the study visit. Participants were required to bring their bottles of IP to each appropriate visit for IP counts for compliance monitoring. Participants could complete participation in the study one month after IP supplementation (Month 2). At the conclusion of the study, participants were no longer eligible to receive IP under this protocol.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 5 | 3
Completed Treatment Completion Visit | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Oral administration of vitamin A palmitate. Vitamin A palmitate: Participants in Cohort 2 were instructed to take 48,000 international unit of investigational product (IP) daily for one month. Participants in Cohort 1 may enroll into Cohort 2 as long as their last intake of vitamin A palmitate was greater than two months prior to their enrollment into Cohort 2. At Baseline, a one month supply of IP was dispensed to the participant during the study visit. Participants were required to bring their bottles of IP to each appropriate visit for IP counts for compliance monitoring. Participants could complete participation in the study one month after IP supplementation (Month 2). At the conclusion of the study, participants were no longer eligible to receive IP under this protocol.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 5 | 3 | 8
Age, Continuous [Median (Standard Deviation); unit: years] | 78.0 (4.74) | 80.0 (7.00) | 78.8 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
Dark Adaptation Rod Intercept Time [Mean (Standard Deviation); unit: minutes] — Baseline measurement of dark adaptation rod intercept time (RIT) in the study eye.
  minutes | 25.12 (10.755) | 20.03 (6.793) | 23.21 (9.285)
Low Luminance Visual Acuity (LLVA) Total Letters Read [Mean (Standard Deviation); unit: letters read] — Baseline measurement of low luminance visual acuity (LLVA) total letters read in the study eye.
  letters read | 66.8 (16.22) | 56.3 (16.17) | 62.9 (15.95)
Low Luminance Questionnaire (LLQ) Composite Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores; (weighted) subscale scores are averaged to produce a composite score.
  score on a scale | 86.35 (17.521) | 86.79 (11.431) | 86.51 (14.588)
Low Luminance Questionnaire (LLQ) Driving Subscale Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
  score on a scale | 86.00 (20.433) | 68.33 (37.859) | 79.38 (27.050)
Low Luminance Questionnaire (LLQ) Extreme Lighting Subscale Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
  score on a scale | 81.25 (18.880) | 73.96 (26.578) | 78.52 (20.488)
Low Luminance Questionnaire (LLQ) Mobility Subscale Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
  score on a scale | 88.33 (16.245) | 96.53 (3.182) | 91.41 (13.102)
Low Luminance Questionnaire (LLQ) Emotional Distress Subscale Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
  score on a scale | 95.00 (8.149) | 97.22 (4.811) | 95.83 (6.774)
Low Luminance Questionnaire (LLQ) General Dim Lighting Subscale Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
  score on a scale | 82.50 (26.087) | 90.28 (2.406) | 85.42 (20.168)
Low Luminance Questionnaire (LLQ) Peripheral Vision Subscale Score [Mean (Standard Deviation); unit: score on a scale] — Low luminance questionnaire (LLQ) is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
  score on a scale | 85.00 (22.361) | 94.44 (9.623) | 88.54 (18.332)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dark Adaptation Rod Intercept Time (RIT) From Baseline in the Study Eye at the Treatment Completion Visit (Month 2 for Cohort 1 and Month 1 for Cohort 2)
Description: The mean change in rod intercept time (RIT) in the study eye at the treatment completion visit from baseline was descriptively summarized and assessed using a Student's paired t-test at a two-sided Type I error rate of 5%.
Time Frame: Baseline to Month 2 for Cohort 1 and Baseline to Month 1 for Cohort 2
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
Minutes
  Baseline Visit | 25.12 (10.755) | 20.03 (6.793)
  Treatment Completion Visit | 22.58 (8.219) | 19.77 (7.753)
  Change from Baseline at the Treatment Completion Visit | -2.54 (4.322) | -0.27 (1.767)
Statistical Analysis 1: Comparison: Cohort 1; Analysis: Student's paired t-test on study eyes alone at a two-sided Type I error rate of 5%. Null hypothesis: the mean RIT at Baseline = the mean RIT at the treatment completion visit (Month 2 for Cohort 1); Test type: Superiority; p = 0.259, Student's paired t-test — Result of statistical analyses were considered significant if the p-value from the two-sided test was <0.05. No adjustments for multiplicity were made; Mean Difference (Final Values) = -2.54, 95% CI 2-sided [-7.91 to 2.83] — The estimate was the difference in mean change in RIT between baseline and the treatment completion visit
Statistical Analysis 2: Comparison: Cohort 2; Analysis: Student's paired t-test on study eyes alone at a two-sided Type I error rate of 5%. Null hypothesis: the mean RIT at Baseline = the mean RIT at the treatment completion visit (Month 1 for Cohort 2); Test type: Superiority; p = 0.818, Student's paired t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-4.66 to 4.12] — The estimate was the difference in mean change in RIT between baseline and the treatment completion visit

2. Secondary Outcome: Change in Dark Adaptation Rod Intercept Time (RIT) From Baseline in the Study Eye at the Post-Treatment Follow-Up Visit (Month 3 for Cohort 1 and Month 2 for Cohort 2).
Description: The mean change in rod intercept time (RIT) in the study eye at the post-treatment follow-up visit from baseline was descriptively summarized and assessed using a Student's paired t-test at a two-sided Type I error rate of 5%.
Time Frame: Baseline to Month 3 for Cohort 1 and Baseline to Month 2 for Cohort 2
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
minutes
  Baseline Visit | 25.12 (10.755) | 20.03 (6.793)
  Post-Treatment Follow-Up Visit | 21.56 (6.271) | 23.27 (12.847)
  Change from Baseline at the Post-Treatment Follow-Up Visit | -3.56 (7.793) | 3.23 (6.512)
Statistical Analysis 1: Comparison: Cohort 1; Analysis: Student's paired t-test on study eyes alone at a two-sided Type I error rate of 5%. Null hypothesis: the mean RIT at Baseline = the mean RIT at the post-treatment follow-up visit (Month 3 for Cohort 1); Test type: Superiority; p = 0.365, Student's paired t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.56, 95% CI 2-sided [-13.24 to 6.12] — The estimate was the difference in mean change in RIT between baseline and the post-treatment follow-up visit
Statistical Analysis 2: Comparison: Cohort 2; Analysis: Student's paired t-test on study eyes alone at a two-sided Type I error rate of 5%. Null hypothesis: the mean RIT at Baseline = the mean RIT at the post-treatment follow-up visit (Month 2 for Cohort 2); Test type: Superiority; p = 0.480, Student's paired t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.23, 95% CI 2-sided [-12.94 to 19.41] — The estimate was the difference in mean change in RIT between baseline and the post-treatment follow-up visit

3. Secondary Outcome: Change in Low Luminance Visual Acuity (LLVA) From Baseline in the Study Eye at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance visual acuity (LLVA) in the study eye from baseline at the treatment completion and post-treatment follow-up visits were descriptively summarized.
Time Frame: Treatment Completion Visit: Month 2 for Cohort 1 and Month 1 for Cohort 2; Post-Treatment Follow-Up Visit: Month 3 for Cohort 1 and Month 2 for Cohort 2
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: letters read
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
letters read
  Baseline Visit | 66.8 (16.22) | 56.3 (16.17)
  Treatment Completion Visit | 71.6 (11.41) | 59.3 (16.01)
  Change from Baseline at the Treatment Completion Visit | 4.8 (17.31) | 3.0 (1.73)
  Post-Treatment Follow-Up Visit | 69.8 (6.69) | 59.3 (17.01)
  Change from Baseline at the Post-Treatment Follow-Up Visit | 3.0 (14.88) | 3.0 (2.00)

4. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) Composite Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) composite score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores; (weighted) subscale scores are averaged to produce a composite score.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 86.35 (17.521) | 86.79 (11.431)
  Treatment Completion Visit | 87.38 (17.420) | 86.13 (9.958)
  Post-Treatment Follow-Up Visit | 84.83 (19.142) | 88.73 (7.382)
  Change from Baseline at the Treatment Completion Visit | 1.03 (1.087) | -0.66 (2.815)
  Change from Baseline at the Post-Treatment Follow-Up Visit | -1.51 (3.283) | 1.93 (5.435)

5. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) Driving Subscale Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) driving subscale score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 86.00 (20.433) | 68.33 (37.859)
  Treatment Completion Visit | 87.00 (17.889) | 55.00 (36.056)
  Post-Treatment Follow-Up Visit | 84.00 (22.192) | 63.33 (33.292)
  Change from Baseline at the Treatment Completion Visit | 1.00 (8.944) | -13.33 (5.774)
  Change from Baseline at the Post-Treatment Follow-Up Visit | -2.00 (4.472) | -5.00 (5.000)

6. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) Extreme Lighting Subscale Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) extreme lighting subscale score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 81.25 (18.880) | 73.96 (26.578)
  Treatment Completion Visit | 84.38 (20.492) | 77.08 (25.259)
  Post-Treatment Follow-Up Visit | 78.75 (20.420) | 80.83 (12.521)
  Change from Baseline at the Treatment Completion Visit | 3.13 (5.846) | 3.13 (5.413)
  Change from Baseline at the Post-Treatment Follow-Up Visit | -2.50 (6.775) | 6.88 (26.612)

7. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) Mobility Subscale Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) mobility subscale score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 88.33 (16.245) | 96.53 (3.182)
  Treatment Completion Visit | 90.00 (14.006) | 97.22 (2.406)
  Post-Treatment Follow-Up Visit | 88.33 (15.975) | 97.22 (2.406)
  Change from Baseline at the Treatment Completion Visit | 1.67 (2.282) | 0.69 (5.243)
  Change from Baseline at the Post-Treatment Follow-Up Visit | 0.00 (2.946) | 0.69 (5.243)

8. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) Emotional Distress Subscale Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) emotional distress subscale score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 95.00 (8.149) | 97.22 (4.811)
  Treatment Completion Visit | 93.75 (10.825) | 95.14 (4.337)
  Post-Treatment Follow-Up Visit | 93.75 (10.825) | 97.92 (3.608)
  Change from Baseline at the Treatment Completion Visit | -1.25 (2.795) | -2.08 (3.608)
  Change from Baseline at the Post-Treatment Follow-Up Visit | -1.25 (2.795) | 0.69 (1.203)

9. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) General Dim Lighting Subscale Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) general dim lighting subscale score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 82.50 (26.087) | 90.28 (2.406)
  Treatment Completion Visit | 84.17 (24.008) | 95.14 (4.337)
  Post-Treatment Follow-Up Visit | 82.50 (25.069) | 93.06 (6.365)
  Change from Baseline at the Treatment Completion Visit | 1.67 (2.282) | 4.86 (4.337)
  Change from Baseline at the Post-Treatment Follow-Up Visit | 0.00 (2.946) | 2.78 (4.811)

10. Secondary Outcome: Change in Low Luminance Questionnaire (LLQ) Peripheral Vision Subscale Score From Baseline at the Treatment Completion and Post-Treatment Follow-Up Visits
Description: The mean change in low luminance questionnaire (LLQ) peripheral vision subscale score from baseline at the treatment completion and post-treatment completion visits were descriptively summarized. LLQ is a 32-item questionnaire relating to difficulty with visual function in low luminance settings. Questions are scored on a range from 0 (indicative of maximum difficulty) to 100 (indicative of no difficulty) in 25 point increments where higher scores indicate better functioning. Each question is assigned to one of six distinct subscales. Applicable questions are averaged to produce (weighted) subscale scores.
Time Frame: as for outcome 3
Population: Primary Analysis Population: Participants enrolled who received IP through the treatment completion visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 5 | 3
score on a scale
  Baseline Visit | 85.00 (22.361) | 94.44 (9.623)
  Treatment Completion Visit | 85.00 (22.361) | 97.22 (4.811)
  Post-Treatment Follow-Up Visit | 81.67 (25.276) | 100.00 (0.000)
  Change from Baseline at the Treatment Completion Visit | 0.00 (0.000) | 2.78 (4.811)
  Change from Baseline at the Post-Treatment Follow-Up Visit | -3.33 (7.454) | 5.56 (9.623)

ADVERSE EVENTS:
Time Frame: Participants enrolled are assessed for AEs starting at Baseline through study completion (Month 3 for Cohort 1 and Month 2 for Cohort 2).
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 2/5 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=3)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Lacrimal disorder (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostatic mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) — Natural Progression of Disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03478865/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT03478865/SAP_001.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT03478865/ICF_002.pdf